CLINICAL TRIAL: NCT06125496
Title: The Relationship Between Kinesiophobia, Physical Activity and Disability Level and Pain Management in Patients With Chronic Low Back Pain in Genders
Brief Title: Relationship Between Kinesiophobia, Physical Activity and Disability Level and Pain Management in Patients With CLBP
Status: Completed | Type: Observational
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayse Unal, Assoc. Prof., Alanya Alaaddin Keykubat University
Other Study IDs: 60116787-020/92289
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain
Keywords: Pain management; Kinesiophobia; Physical activity; Disability
MeSH Terms: conditions — Low Back Pain; Agnosia; Kinesiophobia; Motor Activity | interventions — Pain Management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female: Forty one females with CLBP between the ages of 20-60 participated in the study. Pain management strategies were determined by Pain Coping Questionnaire (PCQ). Tampa Scale for Kinesiophobia for perception of kinesiophobia, Oswestry Disability Index for disability due to pain and International Physical Activity Questionnaire-Short Form (IPAQ-SF) for the physical activity level were used.
  Interventions: Other: Pain management
- Male: Forty one males with CLBP between the ages of 20-60 participated in the study. Pain management strategies were determined by Pain Coping Questionnaire (PCQ). Tampa Scale for Kinesiophobia for perception of kinesiophobia, Oswestry Disability Index for disability due to pain and International Physical Activity Questionnaire-Short Form (IPAQ-SF) for the physical activity level were used.
  Interventions: Other: Pain management

INTERVENTIONS:
Other: Pain management — Investigation of relationship between kinesiophobia, physical activity and disability level and pain management in patients with CLBP

SUMMARY:
The aim of this study was to examine the relationship between pain management, kinesiophobia, physical activity and disability level in patients with chronic low back pain (CLBP) in different genders. Eighty-two patients with CLBP (42 females, 42 males) between the ages of 20-60 participated in the study. Pain management strategies were determined by Pain Coping Questionnaire (PCQ). Tampa Scale for Kinesiophobia for perception of kinesiophobia, Oswestry Disability Index for disability due to pain and International Physical Activity Questionnaire-Short Form (IPAQ-SF) for the physical activity level were used.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are between 20 and 60 years old,
* Experienced low back pain lasting longer than 3 months, and had no problems with reading, writing, and comprehension were included in the study.

Exclusion Criteria:

* Individuals who underwent surgery for low back pain,
* Had any diagnosed spinal problem,
* Who were pregnant,
* And who had communication problems were not included in the study.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: One hundred twenty-six subjects were invited to participate in the study. The study was completed with the participation of 84 subjects, 42 women and 42 men.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Pain Coping Questionnaire (PCQ) | From 25 December 2019 to 10 November 2021
  The scale assesses how chronic pain patients cope with organic or psychogenic pain. The scale consists of four subdimensions that are self-coping, helplessness, conscious cognitive interventions, and seeking medical help, and 29 items. The self-report scale consists of a 4-point Likert scale (0: never, 3: often).

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | From 25 December 2019 to 10 November 2021
  Subjects were asked to mark the severity of pain on a 10-cm line. The lowest point indicated the least severity of pain, and the highest point indicated the maximum pain value.
Oswestry Disability Index (ODI) | From 25 December 2019 to 10 November 2021
  It consists of 10 items measuring the severity of pain, personal care, lifting, walking, sitting, standing, social life, sleeping, traveling, and degree of pain. Each item is scored between 0-5. The higher the total score, the higher the degree of disability. The maximum score is 50 points.
Tampa Scale of Kinesiophobia (TSK) | From 25 December 2019 to 10 November 2021
  The scale is scored between 17 and 68 using a 4-point Likert type scale scoring system. A high score on the scale indicates a high level of kinesiophobia.
International Physical Activity Questionnaire-Short Form (IPAQ -SF) | From 25 December 2019 to 10 November 2021
  The questionnaire provides information on time spent walking, moderate to vigorous activity, and vigorous activity. Time spent sitting is included as a separate question. The total score calculation includes the sum of time (minutes) and frequency (days) of walking, moderate activity, and vigorous activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Ünal, Assoc. Prof, Principal Investigator — Alanya Alaaddin Keykubat University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No